CLINICAL TRIAL: NCT01598727
Title: A Phase I Feasibility Study of Intra-operative Near Infra-red Fluorescent Imaging in Thyroid/Parathyroid Surgery With the Fluobeam(TM) System of Fluoptics
Brief Title: Near Infrared Fluorescent Imaging in Thyroid and Parathyroid Surgery With the Fluobeam(TM) System of Fluoptics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Fluoptics Ltd, Grenoble, France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH16019
Record Dates: First submitted 2012-05-03; First posted 2012-05-15 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Primary Hyperparathyroidism
Keywords: parathyroid surgery
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fluobeam(TM) Imaging System (Fluoptics) (Experimental): Single arm observational pilot study
  Interventions: Device: Fluobeam(TM) Imaging System (Fluoptics)

INTERVENTIONS:
Device: Fluobeam(TM) Imaging System (Fluoptics) — Use of 'Fluobeam(TM)' (Fluoptics) as an intraoperative real time fluorescence detection system during surgery

SUMMARY:
Hypothesis: Intraoperative use of near infrared fluorescent imaging technology and detection of Methylene Blue fluorescence will improve outcomes following thyroid and parathyroid surgery.

Aims: The aims of this phase of the study are to determine the feasibility of using near infrared fluorescent technology in the detection of parathyroid tissue and its differentiation from adjacent soft tissue during surgery on parathyroid glands.

Objectives of the phase I study:

1. To familiarise surgical teams with the intraoperative use of the 'Fluobeam(TM)' device (Fluoptics).
2. To understand the patterns (onset, intensity and duration) of fluorescent staining of normal parathyroid glands, thyroid glands and other soft tissue structures encountered during parathyroidectomy.

Further research:

This will be followed by a phase II study during which fluorescent imaging will be used in conjunction with intraoperative incremental dose of IV methylene blue in both thyroid and parathyroid surgery. Phase II will enable us to develop a protocol for the use of a minimum possible dose of MB for the identification of parathyroid glands. This will then be tested in the pilot phase of a randomized clinical trial.

DETAILED DESCRIPTION:
As above

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing parathyroid surgery

Exclusion Criteria:

* patients undergoing re-do procedures
* patients unable to give adequate informed consent
* patients with a history of intolerance or sensitivity to MB
* patients with G6PD deficiency
* patients on serotonin reuptake inhibitors and patients undergoing thoracic exploration
* either alone or in combination with a neck exploration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Determine patterns of fluorescence from soft tissue structures in the neck | 1 Day
  This is a proof of principle study aimed to demonstrate that the patterns of Methylene Blue emitted fluorescence from the parathyroid glands, thyroid glands and other soft tissue structures in the neck such as lymph glands are distinct and can be used to differentiate between them at surgery. The fluorescence from the various structures will be recorded as 'no', 'mild' and 'yes'.

CONTACTS AND LOCATIONS:
Overall Officials: Saba P Balasubramanian, PhD, Principal Investigator — University of Sheffield
Locations (1):
- Department of General Surgery, Sheffield, South Yorkshire, United Kingdom